CLINICAL TRIAL: NCT04551391
Title: Kidney Recovery After Acute Kidney Injury - Longitudinal Study
Acronym: KRAKIL
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Collaborators: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: ss; MR/S01053X/1 (Other Grant/Funding Number: Medical Research Council)
Record Dates: First submitted 2020-03-03; First posted 2020-09-16 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2022-09

CONDITIONS: Acute Kidney Injury; Chronic Kidney Diseases
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Circulating blood concentration of endothelin and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: (i) Adult aged 16 or over; (ii) Ability to provide informed consent; (iii) Diagnosis of AKI determined as:
  * Previous (within 3 years) eGFR >45 mL/min/1.73m2 OR no history of kidney disease if no recent (within 3 years) blood results available AND
  * Elevated creatinine over 1.5 x previous result OR over 150 μmol/L if no previous value AND
  * Increasing creatinine >= 27μmol/L above index value within 48 hours
  Interventions: Other: Blood and urine sampling
- Control: (i) Adult aged 16 or over; (ii) Ability to provide informed consent; (iii) Admitted to hospital without AKI: (eGFR > 60).
  This group will be recruited contemporaneously with, and matched to, AKI participants by:
  1. Age (± 5 years)
  2. Sex
  3. AKI aetiology (ischaemic, infected, nephrotoxic) 4 (i) History of diabetes or not AND/OR (ii) History of cardiovascular disease or not
  Interventions: Other: Blood and urine sampling

INTERVENTIONS:
Other: Blood and urine sampling — Retinal OCT is a novel, non-invasive method for cross-sectionally imaging the eye's retina and choroid
  Other Names: retinal opticla coherence tomography

SUMMARY:
The endothelin (ET) system is an active target in human Acute Kidney Injury (AKI).

Our primary hypothesis is that the circulating blood concentration of ET will be higher in patients with AKI than in matched controls.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a major health problem being both common and costly. It affects ~20% of hospital inpatients and consumes ~1% of the annual NHS budget. AKI occurs following a diverse range of insults, commonly ischaemia-reperfusion injury (IRI) but also sepsis and drug toxicity. Therapies for AKI are currently supportive and short-term mortality remains high, with ~2 million deaths per year worldwide. In those who survive an episode of AKI, 30% are left with chronic kidney disease (CKD). The remaining 70% that recover full renal function are at ~28-fold increased risk of ultimately developing CKD. This risk is even greater in elderly patients. Importantly, CKD is strongly and independently associated with incident cardiovascular disease (CVD), and together these exert a global socioeconomic burden.

The recognition that AKI and CKD are linked is recent and the molecular pathways that control the transition from acute injury to chronic disease are not well defined. Currently, there are no specific treatments that reduce the risk of progressing to CKD after AKI. Thus, there is an unmet need for therapies that will prevent the transition from AKI to CKD and reduce the cardiovascular burden associated with both. Our preliminary investigations (not yet published) in humans and mice suggest that AKI causes sustained activation of the endothelin (ET) system to the long-term detriment of renal and systemic haemodynamic function. These pilot data form the basis of our project that seeks to determine whether the ET system is active in patients with AKI and, thus, represents a potential target for therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

(i) Adult aged 16 or over; (ii) Ability to provide informed consent; (iii) Diagnosis of AKI determined as:

* Previous (within 3 years) eGFR >45 mL/min/1.73m2 OR no history of kidney disease if no recent (within 3 years) blood results available AND
* Elevated creatinine over 1.5 x previous result OR over 150 μmol/L if no previous value AND
* Increasing creatinine >= 27μmol/L above index value within 48 hours

The control group (N=50) inclusion criteria are:

(i) Adult aged 16 or over; (ii) Ability to provide informed consent; (iii) Admitted to hospital without AKI: (eGFR > 60)

This group will be recruited contemporaneously with, and matched to, AKI participants by:

1. Age (± 5 years)
2. Sex
3. AKI aetiology (ischaemic, infected, nephrotoxic) 4 (i) History of diabetes or not AND/OR (ii) History of cardiovascular disease or not

Exclusion Criteria:

1. Inability to provide informed consent
2. Prisoners
3. Pregnancy or breast feeding
4. Evidence of CKD

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: (i) Adult aged 16 or over; (ii) Ability to provide informed consent; (iii) Diagnosis of AKI
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
To primary outcome aims to measure whether circulating ET is higher in patients with AKI than in matched controls. | 3 years
  as above

SECONDARY OUTCOMES:
The secondary outcome aims to measure differences in urine ET between patients with AKI and matched controls AKI patients that do not fully recover renal function within 90 days will have the highest concentrations of blood and urine ET. | 3 YEARS
  as above

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided